CLINICAL TRIAL: NCT05797051
Title: Application of Hyperspectral Imaging in the Diagnosis of Glomerular Diseases
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Qianfoshan Hospital (Other)
Responsible Party: Principal Investigator, Zunsong Wang, Qianfo Mountain Hospital of Shandong Province, Qianfoshan Hospital
Other Study IDs: liquid biopsy-glomerulopathy
Record Dates: First submitted 2023-03-18; First posted 2023-04-04 (Actual); Last update posted 2023-05-03 (Actual); Status verified 2023-04

CONDITIONS: Glomerulonephritis, IGA; Glomerulonephritis, Membranous; Diabetic Nephropathies; Nephrosis, Lipoid; Hyperspectral Imaging
MeSH Terms: conditions — Glomerulonephritis, IGA; Glomerulonephritis, Membranous; Diabetic Nephropathies; Nephrosis, Lipoid

STUDY DESIGN:
Observational Model: Other | Time Perspective: Other
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (4):
- diabetic nephropathy: Urine samples were collected from patients with IgA nephropathy, idiopathic membranous nephropathy, diabetic nephropathy and minimal change nephropathy. The samples were centrifuged and frozen in a refrigerator at -80 degrees Celsius. The images were divided into a training set and a test set at a fixed ratio. The digital images were input into classification models such as one-dimensional convolutional neural network to learn and test. The training set was used for the training and parameter iteration of the artificial intelligence non-invasive fluid diagnosis model, and the test set was used for the recognition and interpretation of the model. The confusion matrix, accuracy and ROC curve were calculated through the interpretation results to evaluate the performance of the model.
  Interventions: Diagnostic Test: Microscopic hyperspectral imaging system
- minimal change nephropathy: Urine samples were collected from patients with IgA nephropathy, idiopathic membranous nephropathy, diabetic nephropathy and minimal change nephropathy. The samples were centrifuged and frozen in a refrigerator at -80 degrees Celsius. The images were divided into a training set and a test set at a fixed ratio. The digital images were input into classification models such as one-dimensional convolutional neural network to learn and test. The training set was used for the training and parameter iteration of the artificial intelligence non-invasive fluid diagnosis model, and the test set was used for the recognition and interpretation of the model. The confusion matrix, accuracy and ROC curve were calculated through the interpretation results to evaluate the performance of the model.
  Interventions: Diagnostic Test: Microscopic hyperspectral imaging system
- IgA nephropathy: Urine samples were collected from patients with IgA nephropathy, idiopathic membranous nephropathy, diabetic nephropathy and minimal change nephropathy. The samples were centrifuged and frozen in a refrigerator at -80 degrees Celsius. The images were divided into a training set and a test set at a fixed ratio. The digital images were input into classification models such as one-dimensional convolutional neural network to learn and test. The training set was used for the training and parameter iteration of the artificial intelligence non-invasive fluid diagnosis model, and the test set was used for the recognition and interpretation of the model. The confusion matrix, accuracy and ROC curve were calculated through the interpretation results to evaluate the performance of the model.
  Interventions: Diagnostic Test: Microscopic hyperspectral imaging system
- idiopathic membranous nephropathy: Urine samples were collected from patients with IgA nephropathy, idiopathic membranous nephropathy, diabetic nephropathy and minimal change nephropathy. The samples were centrifuged and frozen in a refrigerator at -80 degrees Celsius. The images were divided into a training set and a test set at a fixed ratio. The digital images were input into classification models such as one-dimensional convolutional neural network to learn and test. The training set was used for the training and parameter iteration of the artificial intelligence non-invasive fluid diagnosis model, and the test set was used for the recognition and interpretation of the model. The confusion matrix, accuracy and ROC curve were calculated through the interpretation results to evaluate the performance of the model.
  Interventions: Diagnostic Test: Microscopic hyperspectral imaging system

INTERVENTIONS:
Diagnostic Test: Microscopic hyperspectral imaging system — Microscopic hyperspectral imaging system

SUMMARY:
Morning urine samples of patients with IgA nephropathy, idiopathic membranous nephropathy, diabetic nephropathy, and minimal degenerative nephropathy confirmed by renal needle biopsy in our hospital from November 2020 to January 2022 were collected. By scanning the morning urine samples of corresponding patients with microhyperspectral imager, machine learning and deep learning were used to classify microhyperspectral images, and the classification accuracy was greater than 85%. Thus, hyperspectral imaging technology could be used as a non-invasive diagnostic means to assist the diagnosis of glomerular diseases.

ELIGIBILITY:
Inclusion Criteria:

* Over 18 years old;
* Patients with IgA nephropathy, idiopathic membranous nephropathy, diabetic nephropathy, minimal change nephropathy confirmed by renal biopsy;
* Had not received hormone and/or immunosuppressive therapy before renal biopsy;
* Complete clinical data, all signed the "Admission Certificate of Qianfoshan Hospital of Shandong Province", and agreed to use relevant medical information, biological specimen examination and examination results for scientific research.

Exclusion Criteria:

* There are factors causing secondary membranous nephropathy, such as immune diseases (systemic lupus erythematosus), tumors/infections (viral hepatitis), drugs or poisons, etc.;
* Severe infection: fever, cough and expectoration, sore throat, abdominal pain, diarrhea, carbuncle and furuncle and other clinical manifestations of skin and soft tissue infection, blood routine white blood cell count beyond the normal range (10×109/L);
* Severe cardiovascular disease: including chronic heart failure grade 3 or above and various arrhythmias;
* Infectious diseases: active hepatitis, AIDS, syphilis, etc. ;
* Tumor evidence: it has been found that there is a certain tumor or clinical manifestations, tumor markers, etc., suggesting the possibility of tumor.

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with massive proteinuria were diagnosed as IgA nephropathy, idiopathic membranous nephropathy, diabetic nephropathy and minimal change nephropathy by renal biopsy.
Sampling Method: Probability Sample
Enrollment: 80 (Estimated)
Dates: Start 2023-05-30 (Estimated); Primary Completion 2023-08-20 (Estimated); Study Completion 2023-09-20 (Estimated)

PRIMARY OUTCOMES:
Microhyperspectral image of urine specimen | 2023.4-2023.10
  Microhyperspectral images of urine samples from patients with four different glomerular diseases before treatment